CLINICAL TRIAL: NCT06200753
Title: Triage of Patients Presenting Beyond 24 Hours From Last Known Well With Acute Ischemic Stroke Due to Large Vessel Occlusions (TRACK-LVO Late): a TRACK-LVO Registry-linked Cohort
Brief Title: Triage of Patients Presenting Beyond 24 Hours With Acute Ischemic Stroke Due to Large Vessel Occlusions (TRACK-LVO Late)
Acronym: TRACK-LVO Late
Status: Recruiting | Type: Observational
Sponsor: Tianjin Huanhu Hospital (Other)
Responsible Party: Principal Investigator, Ming Wei, Chief Physician, Tianjin Huanhu Hospital
Other Study IDs: TJHH-2023-WM28
Record Dates: First submitted 2023-12-16; First posted 2024-01-11 (Actual); Last update posted 2024-01-11 (Actual); Status verified 2023-12

CONDITIONS: Endovascular Thrombectomy; Large Vessel Occlusion; Acute Ischemic Stroke
Keywords: Acute Ischemic Stroke, Endovascular Therapy,
MeSH Terms: conditions — Ischemic Stroke | interventions — Ischemic Postconditioning

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Endovascular therapy
  Interventions: Procedure: Mechanical Thrombectomy
- Best medical treatment
  Interventions: Procedure: Mechanical Thrombectomy

INTERVENTIONS:
Procedure: Mechanical Thrombectomy — Mechanical Thrombectomy: A stroke treatment method involving the use of a device to extract a blood clot from the blood vessels, restoring blood flow and reducing brain damage.
  Ischemic Post-conditioning: After thrombectomy, a procedure involving inflating and deflating a balloon in situ for four cycles of 2 minutes each, reducing reperfusion injury and minimizing neural damage.
  Selective Hypothermia: Administering cold saline either intra-arterially or within the cerebral sinus to lower brain temperature, mitigating ischemia-induced injury.
  Other Names: Ischemic post-conditioning; Selective Hypohermia

SUMMARY:
The objective of this study is to create a comprehensive, multi-center, TRACK-LVO registry-linked cohort of consecutive patients with acute ischemic stroke (AIS) caused by large vessel occlusions (LVO) and presenting to each participating center beyond 24 hours from last known well, who are treated with either endovascular therapy (EVT) or the best available medical management (BMM).

DETAILED DESCRIPTION:
There is an abundance of evidence demonstrating the efficacy and safety of endovascular therapy (EVT) within 24 hours of stroke onset. However, the potential benefits of EVT beyond this time window remain uncertain. To address this knowledge gap, the investigators established a TRACK-LVO Late linked cohort, specifically designed to investigate the outcomes of EVT in patients with LVO presenting beyond 24 hours from last known well.

This cohort includes patients from the TRACK-LVO registry who received either EVT or best medical treatment (BMT) beyond 24 hours from symptom onset. The cohort focuses on patients with LVO in the anterior circulation, confirmed by magnetic resonance angiography (MRA), computed tomography angiography (CTA), or digital subtraction angiography (DSA) in the EVT group. To maximize the sample size in the BMT group, the investigators also included patients with LVO confirmed using transcranial Doppler and carotid ultrasonography, in addition to the aforementioned imaging modalities.

Consistent with the TRACK-LVO registry, LVO is defined as an occlusion of the intracranial internal carotid artery (ICA) , M1 and/or M2 segments of the middle cerebral artery (MCA), A1 and/or A2 segments of the anterior cerebral artery (ACA), any segments of vertebral artery (VA), basilar artery (BA), or P1 and/or P2 segments of the posterior cerebral artery (PCA).

The investigators collect comprehensive patient information, including baseline demographic profiles, imaging characteristics such as ischemic core volume and FVH-DWI mismatch, CT/MR perfusion parameters, and treatment-related complications, for both EVT and BMT groups. For patients in the EVT group, the investigators also obtained detailed information on the EVT procedure and angiographic images.

By establishing this cohort, the investigators aim to provide high-level evidence to guide the treatment of a subgroup of stroke patients who present beyond the current guideline-recommended time window for EVT. The findings will contribute to determining the superiority of EVT over BMT in ischemic stroke patients with LVO and extended time from symptom onset.

ELIGIBILITY:
Inclusion Criteria:

* Patient admitted from Jan. 1st 2018 to Jan. 1st 2028;
* Presenting beyond 24 hours from last known well;
* Ischemic stroke confirmed by head CT or MRI;
* Large vessel occlusion confirmed by head CTA or MRA: intracranial internal carotid artery (ICA), middle cerebral artery (MCA M1/M2), anterior cerebral artery (ACA A1/A2), basilar artery (BA), vertebral artery (VA), and posterior cerebral artery (PCA P1/P2);
* Patients receiving either endovascular therapy or best medical treatment.

Exclusion Criteria:

• Presence of any forms of cerebral hemorrhage on CT/MR at admission.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Acute stroke patients with large vessel occlusion and presenting beyond 24 hours from last known well
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2018-01-01 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Modified ranking scale (mRS) at 90 days | 90 days
  A 0-6 scale running from perfect health without symptoms to death.
symptomatic intracranial hemorrhage | 72 hours
  any hemorrhagic transformation on subsequent imaging associated with a neurological decline of at least 4 points increase on the NIHSS score

SECONDARY OUTCOMES:
National Institutes of Health Stroke Scale (NIHSS) scores at 90 days | 1, 3, 5 (or discharge), 7 (or discharge) and 90 days
  The NIHSS is composed of 11 items, each of which scores a specific ability between a 0 and 4. For each item, a score of 0 typically indicates normal function in that specific ability, while a higher score is indicative of some level of impairment. The individual scores from each item are summed in order to calculate a patient's total NIHSS score. The maximum possible score is 42, with the minimum score being a 0.
Occurrence of periprocedural complications | 72 hours
  Periprocedural complications include any intracranial hemorrhage, cerebral edema, brain herniation and pneumonia.
EuroQol five dimensions questionnaire (EQ-5D) | 1 year
  The EQ-5D comprises five questions on mobility, self care, pain, usual activities, and psychological status with three possible answers for each item (1=no problem, 2=moderate problem, 3=severe problem). A summary index with a maximum score of 1 can be derived from these five dimensions by conversion with a table of scores. The maximum score of 1 indicates the best health state, by contrast with the scores of individual questions, where higher scores indicate more severe or frequent problems.

CONTACTS AND LOCATIONS:
Locations (1):
- Tianjin Huanhu Hospital, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: No